CLINICAL TRIAL: NCT02010970
Title: A Phase I, Single-center, Open-label, 3-group, Fixed-sequence Study to Assess the Effect of Itraconazole, a Potent CYP3A4 Inhibitor, or Diltiazem, a Moderate CYP3A4 Inhibitor, on the Pharmacokinetics of AZD3293 and the Effects of AZD3293 on the Pharmacokinetics of Midazolam, a CYP3A4/CYP3A5 Substrate, in Healthy Young Male and Female Volunteers
Brief Title: A Phase I Study in Healthy Volunteers to Assess the Effect of Cytochrome3A4 (CYP3A4) Inhibitors (Diltiazem and Itraconazole) on the Pharmacokinetics (PK) of AZD3293 and the Effects of AZD3293 on the Pharmacokinetics of Midazolam, a Cytochrome 3A4 and Cytochrome 3A5 (CYP3A4/CYP3A5) Substrate
Acronym: AZD3293DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D5010C00004
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Volunteers; Pharmacologic Action
Keywords: phase I; healthy volunteers; AZD3293; itraconazole; diltiazem; medazolam; drug interactions; Pharmacokinetics
MeSH Terms: interventions — Calcium Channel Blockers; Benzodiazepines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 AZD3293-itraconazole (Experimental): Subjects from Group 1 will receive a single dose of AZD3293 as an oral solution on Day 1 . In Group 1, itraconazole will be administered orally twice daily starting on Day 5 for 9 consecutive days (Days 5 to 13). On Day 8, a single dose of AZD3293 will be coadministered as an oral solution after the morning dose of itraconazole. Group 1 subjects will be discharged on Day 14.
  Interventions: Drug: Group 1 AZD3293; Drug: Group 1 Itraconazole
- Group 2 AZD3293-diltiazem (Experimental): Subjects from Group 2 will receive a single dose of AZD3293 as an oral solution on Day 1 . In Group 2, diltiazem will be administered orally once daily starting on Day 5, for 9 consecutive days (Days 5 to 13). On Day 8, a single dose of AZD3293 will be coadministered as an oral solution after the diltiazem dose. Group 2 subjects will be discharged on Day 14.
  Interventions: Drug: Group 2 AZD3293; Drug: Group 2 Diltiazem
- Group 3 AZD3293-midazolam (Experimental): Subjects from Group 3 will receive a single dose of midazolam on Day 1 . AZD3293 will be administered as an oral solution once daily starting on Day 2 for 9 consecutive days (Days 2 to 10) followed by a 7 day wash-out period. On Day 8 and Day 17 a single dose of midazolam will be administered. Group 3 subjects will be discharged on Day 18
  Interventions: Drug: Group 3 AZD3293; Drug: Group 3 Midazolam

INTERVENTIONS:
Drug: Group 1 AZD3293 — AZD3293 oral solution
  Other Names: beta secretase inhibitor
  Arms: Group 1 AZD3293-itraconazole
Drug: Group 2 AZD3293 — AZD3293 oral solution
  Other Names: beta secretase inhibitor
  Arms: Group 2 AZD3293-diltiazem
Drug: Group 3 AZD3293 — AZD3293 oral solution
  Other Names: beta secretase inhibitor
  Arms: Group 3 AZD3293-midazolam
Drug: Group 1 Itraconazole — itraconazole capsule
  Other Names: azole antifungal
  Arms: Group 1 AZD3293-itraconazole
Drug: Group 2 Diltiazem — Diltiazem ER tablet
  Other Names: calcium channel blocker
  Arms: Group 2 AZD3293-diltiazem
Drug: Group 3 Midazolam — midazolam syrup
  Other Names: benzodiazepine
  Arms: Group 3 AZD3293-midazolam

SUMMARY:
This study is a single-center, open-label, 3-group, fixed-sequence drug-drug interaction study to assess the effect of coadministration of multiple-dose itraconazole or diltiazem on the single-dose PK of AZD3293 and the effects of coadministration of single- and multiple-dose AZD3293 on the single-dose PK of midazolam. The study will also evaluate the safety and tolerability of single and multiple oral doses of AZD3293, alone and in combination with itraconazole, diltiazem, and midazolam in healthy young subjects.AZD3293 is being developed for the treatment of Alzheimer's disease

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written, and dated informed consent prior to any study-specific procedures Male and nonfertile female healthy subjects, aged 18 to 55 years at the time of consent
* Body weight ≥50 to ≤100 kg and body mass index (BMI) ≥19 to ≤30 kg/m2
* Clinically normal findings on physical examination in relation to age, as judged by the Investigator
* Male healthy subjects must be willing to use barrier contraception, ie, condoms, even if their partners are post-menopausal, surgically sterile, or using accepted contraceptive methods, from the first day of dosing until 3 months after the last dose of investigational product (IP)

Exclusion Criteria:

* Participation in any prior study of AZD3293
* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may put the subject at risk because of participation in the study, may influence the results, or may limit the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* History of previous or ongoing psychiatric disease/condition including psychosis, affective disorder, anxiety disorder, borderline state and personality disorder according to the criteria in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV), as assessed by the Mini-International Neuropsychiatric Interview (MINI)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The effect of multiple-dose co-administration of CYP3A4 inhibitors on the single-dose PK of AZD3293 measured by assessment of area under the curve over the time (AUC) and maximum concentration | up to day 13
  In Group 1, serial blood samples for AZD3293 plasma concentrations will be collected from predose to 96 hours after administration of AZD3293 on Day 1 and from predose to 144 hours after study drug administration on Day 8. Sparse blood samples for itraconazole plasma concentrations will be collected at predose (prior to administration of AZD3293) on Day 1 and 2 hours after the morning dose of itraconazole on Day 5 through Day 13. In Group 2, serial blood samples for AZD3293 plasma concentrations will be collected from predose to 96 hours after administration of AZD3293 on Day 1 and from predose to 144 hours after study drug administration on Day 8. Sparse blood samples for diltiazem plasma concentrations will be collected at predose (prior to administration of AZD3293) on Day 1 and 3 hours after diltiazem administration on Day 5 through Day 13.
The effect of multiple-dose AZD3293 administration (including the reversibilityof any of its effects) on the single-dose PK of a CYP3A4/CYP3A5 substrate (midazolam) by assessment of area under the curve over the time (AUC) and maximum concentration | up to day 17
  Serial blood samples for midazolam plasma concentrations will be collected from predose to 24 hours after administration of midazolam on Day 1 and Day 17 and for 48 hours after administration of midazolam on Day 8. Sparse blood samples for AZD3293 plasma concentrations will be collected at predose (prior to administration of midazolam) on Day 1 and 2 hours after AZD3293 administration on Day 2 through Day 10.

SECONDARY OUTCOMES:
Safety profile in terms of Adverse events assessment | from Baseline and up to day 18
Safety and tolerability in terms of lab tests assessment (hematology, chemistry, urinalysis) | from Baseline and up to day 18
Safety and tolerability in terms of vital signs assessment (blood pressure, pulse and body temperature) and physical exams | from baseline and up till day 18
Safety and tolerability by assessing changes in electrocardiogram (ECG) parameters | from Baseline and up to day 18
Safety and tolerability by assessing telemetry records | from baseline and up to day 13
Suicidality mesured by Columbia-Suicide Severity Rating Scale (C-SSRS) | from Baseline and up till day 18

CONTACTS AND LOCATIONS:
Overall Officials: Apinya Vutikullird, DO, Principal Investigator — WCCT Global
Locations (1):
- Research Site, Cypress, California, United States